CLINICAL TRIAL: NCT02504970
Title: Anesthesia Quality Institute National Anesthesia Clinical Outcomes Registry Ongoing
Brief Title: Anesthesia Quality Institute National Anesthesia Clinical Outcomes Registry
Acronym: AQINACOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Anesthesia Quality Institute (Other)
Responsible Party: Sponsor
Other Study IDs: AnesthesiaQI
Record Dates: First submitted 2015-06-24; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Anesthesia
Keywords: Anesthesia; Quality Improvement

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anesthesia Group Type: AQI collects data from anesthesia groups. The groups are classified according to practice type

SUMMARY:
The Anesthesia Quality Institute (AQI) is home to the National Anesthesia Clinical Outcomes Registry (NACOR), a data warehouse that has been designated as a Qualified Clinical Data Registry (QCDR) by the Centers for Medicare and Medicaid Services (CMS) for Physician Quality Reporting System (PQRS) reporting. With 20 million cases and growing, Anesthesia Quality Institute's clinical data provides an evidence-based rational that informs treatment choices and helps control treatment costs.

National Anesthesia Clinical Outcomes Registry is intended for all anesthesia providers caring for patients. The registry provides participating providers with:

Custom continuous performance monitors Performance gap analysis and patient outlier identification Access to improvement interventions to close performance gaps including patient care management tools, targeted education, resources and other evidence based interventions Registry and peer-to-peer benchmarks

DETAILED DESCRIPTION:
The Anesthesia Quality Institute is home to the National Anesthesia Clinical Outcomes Registry , a data warehouse that has been designated as a Qualified Clinical Data Registry by the Centers for Medicare and Medicaid Services for Physician Quality Reporting System reporting. With 20 million cases and growing, Anesthesia Quality Institute's clinical data provides an evidence-based rational that informs treatment choices and helps control treatment costs.

National Anesthesia Clinical Outcomes Registry is intended for all anesthesia providers caring for patients. The registry provides participating providers with:

Custom continuous performance monitors Performance gap analysis and patient outlier identification Access to improvement interventions to close performance gaps including patient care management tools, targeted education, resources and other evidence based interventions Registry and peer-to-peer benchmarks

Performance

Participants have unlimited access to National Anesthesia Clinical Outcomes Registry to identify opportunities to improve anesthesia clinical care. Reports allow participants to immediately identify gaps in specific quality measures and focus efforts to close those gaps. Performance tracking reports capture trends over time and help measure improvements in quality care. National Anesthesia Clinical Outcomes Registry also provides participants with access to national benchmarking reports.

Patient Outliers

National Anesthesia Clinical Outcomes Registry participants can also improve care by reviewing performance results across their patient population. This information helps to address clinical gaps in a timely manner. Consider and choose interventions that can lead to sustainable practice improvement for your aggregate performance, which can help reduce the number of patient outliers in the future.

Improvement

National Anesthesia Clinical Outcomes Registry identifies possible interventions for improvement based on clinical quality gaps found through calculating selected data. Data can be used to review performance and determine quickly the impact of an improvement intervention. Results are presented graphically to identify trends in performance.

National Anesthesia Clinical Outcomes Registry is approved by Centers for Medicare and Medicaid Services as a Qualified Clinical Data Registry . A Qualified Clinical Data Registry is a registry comprised of Physician Quality Reporting System (PQRS) and/or non Physician Quality Reporting System-approved measures which qualifies as a Centers for Medicare and Medicaid Services-approved reporting tool for Physician Quality Reporting System. Previously, physician anesthesiologists were limited to reporting three measures to Physician Quality Reporting System. National Anesthesia Clinical Outcomes Registry has more than a dozen additional anesthesia-related measure--helping eligible professionals satisfactorily report on outcomes that matter to them and their patients, and more easily meet Physician Quality Reporting System requirements.

Qualified Clinical Data Registry reporting services are included in American Society of Anesthesiologists (ASA) membership, and all Eligible Professionals may participate through American Society of Anesthesiologists membership. Non-member physicians and non-physicians must pay additional fees. All eligible professionals using Qualified Clinical Data Registry reporting services must be a member of National Anesthesia Clinical Outcomes Registry.

Steps for becoming a National Anesthesia Clinical Outcomes Registry participant

National Anesthesia Clinical Outcomes Registry participants range from pen-and-paper anesthesiology practices to the most wired academic centers. You do not need an AIMS system or electronic health records to participate. Anesthesia Quality Institute will help facilitate the contribution of desired data.

National Anesthesia Clinical Outcomes Registry allows for close collaboration between Anesthesia Quality Institute, individual providers and healthcare technology vendors. Roles are defined as follows:

Anesthesia Quality Institute Key Roles

Define data and outcomes collected in National Anesthesia Clinical Outcomes Registry Provide unifying definitions and templates Contract with individual practices and hospitals to exchange data Report collected data

Individual Anesthesia Practices, Hospitals and Providers Key Roles

Provide data to National Anesthesia Clinical Outcomes Registry Use reports to improve patient care to meet various local, state and federal regulatory requirements

Vendors of Anesthesia Information Technology Key Roes

Facilitate National Anesthesia Clinical Outcomes Registry through reporting work with individuals; vendors that provide formatted data for contribution to National Anesthesia Clinical Outcomes Registry will be listed as Anesthesia Quality Institute Preferred Vendors

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing an anesthetic

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing an anesthetic.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-10; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Patient Centered Outcomes questionnaire | up to 30 days
  Data is collected on a questionnaire completed by the anesthesia provider and submitted to the Anesthesia Quality Institute.

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesia Quality Institute, Schaumburg, Illinois, United States